CLINICAL TRIAL: NCT01338142
Title: A Randomised, Double-Blind, Crossover Bioavailability Study Comparing Amorphous Calcium Carbonate (Acc) Versus Crystalline Calcium Carbonate (Ccc) Using Stable Calcium Isotopes In Postmenopausal Women
Brief Title: Amorphous Calcium Carbonate (Acc) Versus Crystalline Calcium Carbonate (Ccc) Using Stable Calcium Isotopes In Postmenopausal Women
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Amorphical Ltd. (Industry)
Responsible Party: Galit Shaltiel-Gold, Ph.D, Amorphical Ltd. Israel
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TASMC-10-NV-571-CTIL
Record Dates: First submitted 2011-04-13; First posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-03

CONDITIONS: Postmenopause
Keywords: postmenopausal; women; absorption; calcium; amorphous calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CCC (Placebo Comparator): Crystalline calcium carbonate (CCC)
  Interventions: Other: CCC
- ACC (Experimental): Amorphous calcium carbonate (ACC)
  Interventions: Other: ACC

INTERVENTIONS:
Other: CCC — 600 mg (2 capsules of 300 mg) for oral use of 480 mg CCC (192 mg elemental calcium) intrinsically labeled with 15 mg 44Ca and 120 mg of inactive filler, sucrose.
  1.5 mg of 42Ca labeled CaCl2 through IV injection
  Arms: CCC
Other: ACC — 600 mg (2 capsules of 300 mg) for oral use containing 600 mg ACC (192 mg elemental calcium) intrinsically labeled with 15 mg 44Ca 1.5 mg of 42Ca labeled CaCl2 through IV injection
  Arms: ACC

SUMMARY:
The study objective is, to evaluate the fractional absorption of calcium from amorphous calcium carbonate (ACC) Vs crystalline calcium carbonate (CCC) dietary supplements in postmenopausal women.

DETAILED DESCRIPTION:
This is a randomized, double-blind, crossover bioavailability study comparing the fractional absorption of calcium from amorphous calcium carbonate (ACC) versus crystalline calcium carbonate (CCC) using stable calcium isotopes in postmenopausal women.

The study is comprised of 15 subjects orally administered immediately after breakfast a 600 mg gelatin capsules containing either 600 mg (2 capsules of 300 mg)of ACC (192 mg elemental calcium) of 480 mg CCC (192 mg elemental calcium), labeled with 15 mg of 44Ca (2 capsules of 300 mg).

Five minutes following the oral administration, each subject will be infused intravenously with 1.5 mg of CaCl2 labeled with 42Ca over 10 min. Over the following 24 h subjects will consume meals that will be selected by the Unit of Clinical Nutrition at Sourasky Medical Center nutritionist on the basis of their food diary and ALL urine excreted during this time should be collected in a designated urine container and returned to the Unit of Clinical Nutrition at Sourasky Medical Center for evaluation. The same protocol as in day 0 with a crossover oral treatment will be performed after 21 day washout period.

Dosing day will be designated "Day 0". Eligible subjects are randomly assigned to one of the study treatments according to the following regimens:

ELIGIBILITY:
INCLUSION CRITERIA

• Absence of menstrual period for 12 months but not more than 5 years, or absence of menstrual period for 6 to 12 months and follicle stimulating factor (FSH) greater than 40 IU/L

1. BMI 18-29 (inclusive)
2. Subjects able to adhere to the visit schedule and protocol requirements and be available to complete the study.
3. Subjects who provide written informed consent to participate in the study.

EXCLUSION CRITERIA

1. Women who, on the basis of a food frequency questionnaire, have an estimated daily calcium intake >1100 mg through combined diet (both supplements and food).
2. Women with vitamin D deficiency < 30 ng/ml
3. Women with hypercalcemia, nephrolithiasis, inflammatory bowel disease, malabsorption, chronic diarrhea, use of antibiotics within the past month, Woman suffering from digestive, hepatic, renal, or inflammatory diseases.
4. Women who take oral steroids, anticonvulsants, bisphosphonates, estrogen compounds, calcitonin, or teriparatide within the past 6 months.
5. Any acute medical situation (e.g. acute infection) within 48 hours of study start, which is considered of significance by the Principal Investigator (PI).
6. Subjects who are non-cooperative or unwilling to sign consent form.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-05 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Mean change in fractional absorption of calcium from amorphous calcium carbonate (ACC) Vs. crystalline calcium carbonate (CCC). | 1 year
  Fractional absorption will be evaluated by measuring 42Ca and 44Ca levels in the urine over 24 hours (the ratio)

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel